CLINICAL TRIAL: NCT03014388
Title: Posterior Maxillary Ridge Augmentation With Sinus Lift Using Mineralized Plasmatic Matrix Versus Autogenous Bone Graft (A Randomized Clinical Trial Comparative Study)
Brief Title: Posterior Maxillary Ridge Augmentation With Sinus Lift Using Mineralized Plasmatic Matrix Versus Autogenous Bone Graft
Acronym: MPM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Refaat Ragab Abu Ellill, Dentist at menistry of health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU MPM
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-12

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autogenous bone graft (Gold Standard). (Experimental): Patients with defective posterior maxillary alveolar ridges requiring implant insertion will have Autogenous bone graft (Gold standard) and to be used for bone augmentation with sinus lift.
  Interventions: Other: autogenous bone
- Mineralized Plasmatic Matrix (MPM) (Experimental): Patients with defective posterior maxillary alveolar ridges requiring implant insertion will receive bone graft using Mineralized plasmatic matrix.
  Interventions: Other: Mineralized plasmatic matrix

INTERVENTIONS:
Other: autogenous bone — Autogenous bone graft (gold standard). sinus lift with autogenous bone.
  Other Names: Autobone
  Arms: Autogenous bone graft (Gold Standard).
Other: Mineralized plasmatic matrix — By using venoud blood from the patient, together with bone graft, a centrifuge will be used to obtain the top layer after centrifuging blood at 3000 RPM.
  Other Names: MPM
  Arms: Mineralized Plasmatic Matrix (MPM)

SUMMARY:
Using growth factors obtained from patient's venous blood mixed with particulate autogenous bone the study compares bone gain by implant with gold standards in sinus Lift procedures for future implant insertion.

DETAILED DESCRIPTION:
To study the effectiveness of MPM in ridge augmentation with implant insertion compared with autogenous bone graft.

-PICO Population(P) : Patients with defective posterior maxillary alveolar ridge. Intervention (I) :Implant placement and ridge augmentation with MPM. Comparator (C) : Autogenous bone graft. Outcome (O) : Patient satisfaction - Implant stability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients systemically free.
2. Patients with posterior maxillary defective ridges indicated for sinus lift procedure.
3. Cases with 5 mm bone height or less are included in the study.
4. Age between 18 and 50 years.
5. Both sexes.
6. Patients physically able to tolerate surgical and restorative procedures.
7. Good oral hygiene.
8. Highly motivated patients.

Exclusion Criteria:

1. Patients allergic to local anesthetic agent.
2. Medium and heavy smokers.
3. Pregnant females.
4. Presence of any pathosis in the pre-implant site.
5. Presence of any mucosal disease.
6. History of oral radiotherapy.
7. History of prolonged steroids use.
8. Psychological disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction regarding aesthetic results will be measured using questionnaire. | 9 months
  outcome will be measure using questionnaire.

SECONDARY OUTCOMES:
Stability of dental implants. | 5 months
  will be measured using OSTELL Device.

CONTACTS AND LOCATIONS:
Overall Officials: Cairo University CBE, Principal Investigator — Cairo University - Ethics Committee.

IPD SHARING:
Plan to Share IPD: No
Evaluation of the comparative Effectiveness of MPM Augmentation in posterior maxillary ridge defects with Autogenous bone graft.